CLINICAL TRIAL: NCT01067989
Title: Antiangiogenic Treatment Strategy With Metronomic Chemotherapy Regimen Combined With a Cox-2 Inhibitor and a Bisphosphonate for Patients With Metastatic Breast Cancer
Brief Title: Low-Dose/Metronomic(LDM)Chemotherapy for Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No satisfactory acrual
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, LOVEN DAVID, Oncologist, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0078-09-EMC
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Chemotherapy; Breast Cancer, Metastatic
Keywords: metronomic chemotherapy; anti-angiogenic effect; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Cyclophosphamide; Capecitabine; Methotrexate; Celecoxib; Pamidronate; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Experimental): same treatment for all patients
  Interventions: Drug: Cyclophosphamide, Capecitabine, Methotrexate, Celecoxib, Pamidronate (or Zoledronate)

INTERVENTIONS:
Drug: Cyclophosphamide, Capecitabine, Methotrexate, Celecoxib, Pamidronate (or Zoledronate) — 1. Cyclophosphamide Tab. 50mg, 1x1/day, continuously.
  2. Capecitabine Tab. 500mg, 1+2/day, continuously.
  3. Methotrexate Tab. 2.5mg, 1x2/day, 2 days every week.
  4. Celecoxib Tab. 200mg, 1x2/day, continuously.
  5. Pamidronate I.V. 90mg, every 4 weeks; or Zoledronate I.V. 4mg, every 4 weeks)

SUMMARY:
Low-dose metronomic(LDM)chemotherapy as well as anti-inflammatory agents and bisphosphonates have shown anti-angiogenic properties on tumor vasculature.

This study is meant to test the therapeutic potential of an anti-angiogenic treatment strategy by combining all these agents for metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of infiltrating duct carcinoma of breast.
* Her-2 negative tumors.
* ECOG performance status: 0-1.
* Presence of measurable disease: primary and/or metastatic.
* CBC showing normal values or any toxicity limited to grade I.
* SMA showing liver and renal functions < 1.5 normal values
* previous treatment with an anthracycline and with a taxane is mandatory either as neoadjuvant/adjuvant treatment or for metastatic disease.
* previous treatment by chemotherapy for metastatic disease is allowed (up to three lines, allowing for MTD Capecitabine to be one of them).
* previous treatment by a bisphosphonate is allowed. However,those patients who up to the study had not received any bisphosphonate and those who had received Clodronate- will receive Pamidronate; those who had been under Pamidronate- will receive Zoledronate; those who had been under Zoledronate- will continue with it."
* The patient's signature on the informed consent.

Exclusion Criteria:

* Her-2 neu positive tumor
* Inability to visit the clinic for outpatient treatment and evaluation
* Active/symptomatic brain metastases.
* ECOG performance status: 2-4.
* Presence of Hand -Foot syndrome, at grade > 2.
* CBC with any grade >2 toxicity
* SMA showing liver functions > 1.5 normal values
* SMA showing renal functions > normal values -Current continuous treatment by steroids or by NSAIDs, or by anti- coagulants for "non protocol" reasons.
* presence of exclusively non-measurable disease (I/E: exclusive bone disease with non-representative tumor markers).
* previous radiotherapy to the "only measurable disease".
* pleural or peritoneal effusion that may represent a "third space".
* history of active peptic ulcer.
* symptomatic coronary heart disease.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy by rate of clinical benefit (CB): rate of response (RR) + rate of Stable Disease (SD) | 6 and 12 months

SECONDARY OUTCOMES:
Plasma Levels of angiogenic growth factors | At 4 predetermined time points along treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology unit, Afula, Israel